CLINICAL TRIAL: NCT03063814
Title: Immediate Effects of App-based Versus Personal On-site Instruction on Neuromuscular Activity in Injury Prevention Exercises: Randomized Controlled Trial
Brief Title: Effects of App-based Versus Personal On-site Instruction on Neuromuscular Activity in Injury Prevention Exercises
Acronym: ACL01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: Metropolitan University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACL01
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Musculoskeletal Injury; Injury, Knee
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP (Experimental): In the APP group, a video sequence of each exercise, supported by short written descriptions (in accordance to 'Get set - Train smarter', (9) on how to perform the exercise correctly, was shown to the participants on an iPad. The video-recorded exercises were performed by the same physiotherapist who supervised PHY participants. If required, the participants in the APP group were allowed to watch the video and description several times between trials of the same exercise. The participants approved their own trials when they believed that the exercises had been performed as described.
  Interventions: Behavioral: APP
- PHY (Active Comparator): In PHY, a physiotherapist demonstrated and explained the focus areas of each of the five exercises before the participant performed the exercises. If needed, verbal feedback was given between trials to correct the performance of the exercise. The physiotherapist approved trials that were performed with proper technique.
  Interventions: Behavioral: PHY

INTERVENTIONS:
Behavioral: APP — See arm description
  Arms: APP
Behavioral: PHY — see arm description
  Arms: PHY

SUMMARY:
Therefore, the aim of the present study was to evaluate neuromuscular characteristics observed during a single bout of selected and validated injury preventive exercises instructed by an app (in accordance with 'Get set - Train smarter') versus gold standard instruction, supervision and feedback provided on-site by an expert. The present evaluation targets a population of female football and handball players without any previous exposure to injury prevention training.

ELIGIBILITY:
Inclusion Criteria:

* female handball or football player (≥ 18 years old) competing at sub-elite level (i.e., 2-3 weekly training sessions)

Exclusion Criteria:

* previous traumatic knee injury, lower limb injury at the time of testing and/or previous engagement in injury prevention practices.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Normalized hamstring EMG | 5 minutes after instruction
  Normalized to isometric MVC hamstring muscle EMG amplitude recorded during the exercise.

SECONDARY OUTCOMES:
Normalized quadriceps EMG | 5 minutes after instruction
  Normalized EMG amplitude of the quadriceps muscle recorded during the exercise.
Joint angle | 5 minutes after instruction
  Joint angle during the exercise

CONTACTS AND LOCATIONS:
Overall Officials: Mette K Zebis, PhD, Principal Investigator — Metropolitan University College
Locations (1):
- Hvidovre Hospital, Hivdovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided